CLINICAL TRIAL: NCT06772389
Title: The Effect of Electronic Fetal Monitoring Training Given to Midwifery Students With Peer Education Method on the Knowledge, Skills and Self-Efficacy Levels of the Students
Brief Title: Teaching Electronic Fetal Monitoring to Midwifery Students With Peer Teaching Method
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Melek Şen Aytekin, Research Assistant, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GaziosmanpasaU-EBE-MŞA-01
Record Dates: First submitted 2024-12-23; First posted 2025-01-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Educational Problems
Keywords: midwifery; education; cardiotocography; Clinical Skill; peer group

STUDY DESIGN:
Intervention Model Description: The students included in the study were randomly assigned to Peer Tutoring and Standard Education groups.
Who Masked: Outcomes Assessor
Masking Description: After the data collection process of the study is completed, the data will be transferred to the SPSS program by the researcher. When the data is transferred to SPSS by the researcher, the Peer Tutoring group will be given the code X and the Standard Education group will be given the code Y. The person who will perform the statistical analysis will not know which number is which group. After the analysis is completed, the codes will be given their own names and the results will be evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Education Group (No Intervention): This group received standard training given within the scope of the Prenatal Period I course. A powerpoint presentation consisting of 80 slides was prepared within the scope of this training. The training was given as 2 lessons of 50 minutes each. Powerpoint presentation and "Leopold Maneuver Palpation Model" were used during the training.
- Peer Tutoring Group (Experimental): This group received standard training as part of the Prenatal Period I course. A powerpoint presentation consisting of 80 slides was prepared as part of this training. The training was given as 2 lessons of 50 minutes each. A powerpoint presentation and "Leopold Maneuver Palpation Model" were used during the training. Peer training was given two days after the standard training was completed. During the peer training, the powerpoint presentation and the Leopold Maneuver Palpation Model used in standard training were also used.
  Interventions: Other: Peer Tutoring

INTERVENTIONS:
Other: Peer Tutoring — Peer tutoring is defined as "individuals who are in a similar social group and are not professional teachers helping each other to learn and teach". For peer tutoring, the subject of EFM was grouped under 6 headings. The students in the Peer tutoring group were divided into groups of 6. The researcher explained a heading of the EFM subject to each of these 6 groups. Then, new groups were formed by taking one student from each group. In these new groups, each student explained his/her own subject to his/her peers.
  Arms: Peer Tutoring Group

SUMMARY:
706 / 5.000 The aim of the study is to examine the effects of Electronic Fetal Monitoring (EFM) (a test that evaluates fetal health during pregnancy) training given to midwifery students through peer education method on the knowledge, skills and self-efficacy levels of the students. It is being conducted as an experimental study with a randomized controlled pre-test-post-test design. Students were given standard training on EFM. Students in the peer teaching group were given peer education. Students continue to be evaluated while applying EFM to pregnant women in clinical practice. Personal information form, achievement test for EFM, skill form and Electronic Fetal Monitoring Self-Efficacy Scale were used in the evaluation of the students.

DETAILED DESCRIPTION:
The aim of the study was to examine the effects of Electronic Fetal Monitoring (EFM) training given to midwifery students through peer education method on the knowledge, skill and self-efficacy levels of the students. It is being conducted as an experimental study with a randomized controlled pre-test-post-test design.

The Electronic Fetal Monitoring Achievement Test and Electronic Fetal Monitoring Skill Form to be used within the scope of the study were created in line with the literature and presented to the opinions of experts in the field. The necessary arrangements were made in line with the opinions of expert instructors and the final version of the achievement test and skill form was created. The Electronic Fetal Monitoring Self-Efficacy Scale is a valid and reliable scale developed by researchers in Turkey in 2023.

After the measurement tools were completed, standard training on EFM was given to the 2nd year students of the midwifery department within the scope of the Prenatal Period I course. After the standard training, the students were informed about the research. The students included in the study were provided with the Personal information formi achievement test and Electronic Fetal Monitoring Self-Efficacy Scale for EFM as a pre-test. The students included in the study were randomized and assigned to Peer Tutoring and Standard Education groups. Then, peer education was given to the students in the Peer Tutoring group.

After the peer education was completed, all students began to be evaluated while performing EFM on pregnant women in clinical practice. Students are evaluated with a skill form by the researcher while performing EFM on pregnant women. After the application is completed, students complete the EFM achievement test and Electronic Fetal Monitoring Self-Efficacy Scale as a post-test. Evaluation of students continues in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* volunteers to participate in the study,
* those taking the Prenatal Period-I course for the first time,
* those who have not received any EFM training before,
* those who are second year Midwifery students

Exclusion Criteria:

* Students who are absent on the day the EFM topic is taught.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Electronic Fetal Monitoring Self-Efficacy Scale | It will be used as a pre-test 10 minutes after the standard training. As a post-test, it will be filled out within 30 minutes after students complete the EFM application to pregnant women.
  The scale consists of 32 items on a 4-point Likert scale ranging from "Very sure" to "Not sure". A general score is obtained by summing up all items. A high score indicates that EFM Follow-up self-efficacy is high. The lowest score to be obtained from the scale varies between 32 and the highest score varies between 128. There is no cut-off score for the scale.
Success Test for Electronic Fetal Monitoring Success Test for Electronic Fetal Monitoring | It will be used as a pre-test 10 minutes after the standard training. As a post-test, it will be filled out within 30 minutes after students complete the EFM application to pregnant women.
  Electronic Fetal Monitoring Achievement Test was prepared in accordance with the literature with multiple choice (4 options) questions in order to measure the knowledge, skills and abilities acquired by the students. The opinions of 11 faculty members who are experts in the field of midwifery were taken for the achievement test that was created. The content validity of the Electronic Fetal Monitoring Achievement Test was calculated in accordance with the opinions received from the experts. There are 22 questions in the final version of the achievement test. One point is taken for each question answered correctly and 0 points are taken for each question answered incorrectly. The highest score from the achievement test is 22 and the lowest is 0. The higher the total score from the achievement test, the higher the success towards EFM.
Skill Form for Electronic Fetal Monitoring | The EFM application process takes approximately 30 minutes. Students are monitored through this form throughout the process (approximately 30 minutes).
  The form was used to evaluate the application that students will perform during clinical practice. The form includes sections that include welcoming the pregnant woman, connecting her to EFM, following her up, interpreting the EFM trace, determining risks and interventions. The researcher who observed the form evaluated the students as "did not do it (0): The step was applied incorrectly" and "did (1): The step was done correctly". Opinions were received from 11 midwifery experts for the form. In line with the opinions of the experts, the scope validity of the Skill Form for Electronic Fetal Monitoring was calculated. Necessary arrangements were made in terms of language and expression in line with the expert opinions. The final form consists of 39 items. The highest score that can be obtained from the form is 39 and the lowest score is 0. High scores indicate that the skill for EFM is high.

SECONDARY OUTCOMES:
Personal Information Form | It is filled out as a pre-test 10 minutes after the standard training.
  Personal Information Form Personal Information Form was created by the researcher in line with the literature to determine the socio-demographic characteristics of the students (age, education level, employment status, health insurance, parents' education status, parents' profession, etc.). There are 7 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Ş Aytekin, RA, Principal Investigator — Tokat Gaziosmanpasa Universty
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No